CLINICAL TRIAL: NCT07004920
Title: Adaptation and Validation of a Patient-centered Outcome Scale for People in the Intensive Care Unit (IPOS-ICU)
Acronym: IPOS-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: King's College London (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-3146; 2025-3146 (Other: Ethics Committee at the Medical Faculty of Heinrich Heine University Düsseldorf)
Record Dates: First submitted 2025-04-30; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-01

CONDITIONS: Intensive Care Unit Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IPOS-ICU — This is a prospective observational study. Health care providers will be asked to will out the IPOS-ICU for patients in the intensive care unit.

SUMMARY:
The focus of intensive care is on survival and the prolongation of life. The care of organ systems takes priority and is assessed through screening tools such as the Sequential Organ Failure Assessment (SOFA) score, which evaluates clinical and laboratory factors associated with prognosis. Despite advancements in modern intensive care, the hospital mortality rate for mechanically ventilated patients in 2022 was approximately 43%. Even for survivors of intensive care, post-intensive care syndrome poses a significant burden on quality of life.

Although intensive care and palliative care often appear to be contradictory, clinical overlap between these populations is common, with both experiencing physical, psychosocial, and spiritual challenges that frequently require input from specialized teams. Nevertheless, palliative care remains underrepresented in German intensive care units (ICUs), with only 1.4% of ICU patients on prolonged mechanical ventilation receiving specialist palliative care. Therefore, the identification of patients in need of palliative care and the reduction of barriers such as limited resources and varying clinician attitudes must be addressed. This necessitates a robust tool for measuring and assessing palliative care needs specifically in ICU patients, enabling the implementation of interventions aimed at minimizing the burden on patients, families, and treating clinicians, as well as guiding appropriate allocation of healthcare resources.

The Integrated Palliative Care Outcome Scale (IPOS) questionnaire was developed as a patient-centered measurement instrument from a palliative care perspective. IPOS enables the assessment of symptoms and needs from the viewpoint of patients and their families. For patients with COVID-19, an adapted version-IPOS-COV-was developed, wherein healthcare personnel assess patient symptoms and needs. However, no existing instrument comprehensively captures the physical, psychosocial, and spiritual needs of ICU patients and their families from a palliative care perspective. Such a tool could facilitate both the identification of patients requiring palliative care and serve as an endpoint for evaluating the effectiveness of palliative care interventions in ICU settings, including post-discharge outcomes related to post-intensive care syndrome affecting both patients and families.

The underlying hypothesis is that a patient-centered measurement instrument addressing physical, psychosocial, and spiritual needs from a palliative care perspective for ICU patients can be developed and validated based on the IPOS. Additionally, demographic data, clinical course, ICU interventions (e.g., mechanical ventilation, dialysis, palliative care consultations, family discussions, and therapy goal limitations), as well as SOFA scores and Palliative Phase of Illness (PPoI) classifications at the time of IPOS-ICU assessment, will be collected. It is hypothesized that IPOS-ICU scores will correlate with disease severity (as measured by SOFA and PPoI) and poor ICU outcomes, including length of stay, mortality, and discharge location. Furthermore, it is hypothesized that interventions such as palliative care consultations will be associated with lower IPOS-ICU scores. In the first phase of the study, an international and multiprofessional expert panel with experience in both intensive and palliative care will adapt the IPOS questionnaire for ICU patients, resulting in the development of the IPOS-ICU. The following modification strategies will be applied: rewording, removal, addition of items, adjustment of recall periods, and inclusion of a "cannot assess" response option. Online meetings will be conducted with representatives from Germany, Switzerland, the United Kingdom, the Czech Republic, and the United States. A larger review team will then evaluate the adapted version, and an informal "comfort consultation" will be conducted in ICU settings to ensure that the IPOS-ICU is considered appropriate and acceptable by ICU staff. Following adaptation, the validation phase will be conducted using a multicenter design. After obtaining informed consent from study participants, the IPOS-ICU will be administered at designated time points identified during the adaptation process. ICU staff (including at least one nursing professional and one medical professional) will complete the IPOS-ICU. The questionnaire will include an assessment of the PPoI (categorized as stable, unstable, deteriorating, dying, or deceased), and a free-text field for recording the estimated number of hours spent with the patient. Electronic Case Report Forms will capture demographic data, SOFA scores, treatment details, and outcomes following ICU discharge, all extracted from medical records. This study holds significant relevance by addressing the gap between the identification of palliative care needs and the actual implementation and evaluation of palliative care in ICU settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients
* written informed consent from patient or health-care proxy

Exclusion Criteria:

* age < 18 years
* Language barrier (communication in German/local language or English not possible).
* ICU discharge 24h after admission
* no written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged above 18 years in the ICU will be screened for inclusion.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
IPOS-ICU total score | during the intervention
  The primary outcome is the IPOS-ICU and its descriptive analysis. Each of the IPOS-ICU items will have the following units of measure: Not at all (0), Slightly (1), Moderately (2), Severely (3), Overwhelmingly (4), Cannot assess (e.g. unconscious). The investigators will calculate the total score of the IPOS-ICU at each time point of assessment.

SECONDARY OUTCOMES:
Number of positive IPOS-ICU items | during the intervention
  The investigators will determine the incidence of total positive (items with unit >1) items and the total of cannot assess answers.
Palliative Phase of Illness (PPoI) | during the intervention
  Categories: stable, unstable, deteriorating, dying, or deceased
SOFA score | during the intervention
  The Sequential Organ Failure Assessment (SOFA) score is a clinical tool used to assess the extent of a patient's organ dysfunction in the ICU. It evaluates six organ systems: respiratory, cardiovascular, hepatic, coagulation, renal, and neurological. Each system is scored from 0 (normal function) to 4 (most severe dysfunction), resulting in a total score ranging from 0 to 24.
Days of mechanical ventilation | immediately after the intervention
  Number of days of invasive mechanical ventilation via either an endotracheal tube or tracheal cannula in the ICU.
Days of ECMO | immediately after the intervention
  Number of days of extracorporeal membrane oxygenation (ECMO, VV (veno-venous), VA (veno-arterial), and VVA (veno-veno-arterial)) in the ICU.
Days of dialysis | immediately after the intervention
  Number of days of renal replacement therapy in the ICU.
ICU length of stay | immediately after the intervention
  Number of days in the ICU.
ICU mortality | immediately after the intervention
  % of patients dying in the ICU.
ICU discharge location | immediately after the intervention
  ICU discharge to the following categories: Hospital unit, other ICU in the hospital, external ICU, skilled nursing facility, rehabilitation unit, palliative care unit, hospice, home, or other.
Functional status at ICU discharge | immediately after the intervention
  Categorized as: fully independent, partially dependent, or fully dependent.
Clinical Frailty Scale (CFS) at ICU discharge | immediately after the intervention
  The Clinical Frailty Scale is a 9-point scale used to assess a patient's level of frailty based on physical fitness and functional status. It ranges from 1 (Very Fit) to 9 (Terminally Ill). Higher scores indicate worse outcomes, representing greater frailty and increased vulnerability to adverse events, including mortality and poor recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No